CLINICAL TRIAL: NCT05589090
Title: Adaptación y evaluación Del Programa transdiagnóstico Super Skills for Life Aplicado Online Para niños Con Problemas Interiorizados
Brief Title: Super Skills for Life Effectiveness in the Online Modality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Principal Investigator, Mireia Orgilés Amorós, Director, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: DPS.MO.01.17
Record Dates: First submitted 2022-10-17; First posted 2022-10-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Depressive Disorder; Depressive Symptoms; Anxiety Disorders; Anxiety Disorders and Symptoms; Mood Disorders; Child Mental Disorder; Emotional Disorder
Keywords: Super Skills for Life; emotional problems; internalizing problems; children; anxiety; depression
MeSH Terms: conditions — Depressive Disorder; Depression; Anxiety Disorders; Mood Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: Study participants who met the inclusion criteria were randomly assigned to the experimental and control groups. The control group did not receive any intervention during the eight-week duration of the program. However, both groups underwent pretest and posttest assessments. Children assigned to the control group will receive the intervention after the 12-month follow-up assessment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Super Skills for Life intervention
  Interventions: Behavioral: Super Skills for Life program
- Wait-list group (No Intervention): Children in this group did not receive any phycological (public or private) intervention during the eight-week duration of the SSL program. They were informed that children in this group will receive the intervention once the follow-up visit is completed.

INTERVENTIONS:
Behavioral: Super Skills for Life program — Children in the experimental group received eight sessions of the Super Skills for Life protocol. The intervention was implemented using a structured manual for the therapist and a workbook for the children [Orgilés, M., Espada, J.P., Ollendick, T.H. & Essau, C. (2022). Programa Super Skills. Manual del aplicador. Elche, ES: Universidad Miguel Hernández]. The intervention was administered via an online virtual platform for eight weeks, with each session lasting approximately one hour.
  Arms: Intervention group

SUMMARY:
The study aims to evaluate the effectiveness of the transdiagnostic program Super Skills for Life (SSL). This protocol targets children aged 8 to 12 with emotional problems (anxiety, depression, low self-esteem, and lack of social skills). SSL consists of eight sessions targeting common risk factors for internalizing disorders such as cognitive distortions, avoidance, emotional management, low self-esteem, social skills deficits, and coping strategies. The present research focuses on assessing the effectiveness of SSL applied online (through a virtual platform).

DETAILED DESCRIPTION:
After selecting the children based on the online questionnaires completed by the parents (preintervention assessment) and inclusion/exclusion criteria, they were randomly allocated to the conditions of the intervention group and the wait-list control group. Parents and children from both groups completed the same measures at baseline, post-treatment, and 12 months follow-up. Children in the experimental group received the SSL program by the virtual platform.

The objective of the study is to evaluate the benefits of the Super Skills for Life protocol applied online. For this purpose, the researchers will test to what extent the experimental group decreases its anxiety symptoms, anxiety impairment, depressive symptoms, behavioral problems, hyperactivity/inattention, and peer relationship problems, and increase its self-esteem and prosocial behaviors, compared to the control group.

In conclusion, the purpose of the study is to explore whether SSL implemented online can be a cost-effective psychological intervention to prevent emotional problems in Spanish children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-12
* Presenting subclinical symptoms of emotional problems (anxiety, depression)
* Speaking, reading, writing, and understanding Spanish.
* Not receiving psychological or pharmacological treatment for emotional and/or behavioral problems

Exclusion Criteria:

* Had a psychiatric diagnosis already established
* Presenting a severe developmental disorder (intellectual disability, autism spectrum disorder, etc).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline depression symptoms to immediately after the intervention | 1 year after the intervention
  Measured by the Mood and Feelings Questionnaire (MFQ-C; short version), a screening tool for depression in children aged 6-17 years. Children must report their feelings and behaviors over the previous 2 weeks. The sum of all items provides a total measure of depression (score range: 0-26), and the higher this score is, the more severe the symptoms are.
Depression symptoms at 1 year | 1 year after the intervention
  Measured by the Mood and Feelings Questionnaire (MFQ-C; short version), a screening tool for depression in children aged 6-17 years. Children must report their feelings and behaviors over the previous 2 weeks. The sum of all items provides a total measure of depression (score range: 0-26), and the higher this score is, the more severe the symptoms are.
Change from baseline parent-reported depression to immediately after the intervention | baseline and immediately after the intervention
  Measured by the Mood and Feelings Questionnaire (MFQ-P; short version), a screening tool for depression in children aged 6-17 years. Parents must inform about their children's feelings and behaviors over the previous 2 weeks. The sum of all items provides a total measure of depression (score range: 0-26), and the higher this score is, the more severe the symptoms are.
Parent-reported depression at 1 year | 1 year after the intervention
  Measured by the Mood and Feelings Questionnaire (MFQ-P; short version), a screening tool for depression in children aged 6-17 years. Parents must inform about their children's feelings and behaviors over the previous 2 weeks. The sum of all items provides a total measure of depression (score range: 0-26), and the higher this score is, the more severe the symptoms are.
Change from baseline children's reported anxiety symptoms to immediately after the intervention | baseline and immediately after the intervention
  Measured by Spence Children's Anxiety Scale Child Report (SCAS; short version). SCAS measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety, and specific fears). This yields a minimum possible score of 0 and a maximum possible score of 24. Higher scores indicate greater severity of symptoms
Change from baseline parent-reported anxiety symptoms to immediately after the intervention | baseline and immediately after the intervention
  Measured by Spence Children's Anxiety Scale Parent Report (SCAS-P; short version). SCAS-P measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety, and specific fears). This yields a minimum possible score of 0 and a maximum possible score of 24. Higher scores indicate greater severity of symptoms.
Children's reported anxiety symptoms at 1 year | 1 year after the intervention
  Measured by Spence Children's Anxiety Scale Child Report (SCAS; short version). SCAS measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety, and specific fears). This yields a minimum possible score of 0 and a maximum possible score of 24. Higher scores indicate greater severity of symptoms
Parent-reported anxiety at 1 year | 1 year after the intervention
  Measured by Spence Children's Anxiety Scale Parent Report (SCAS-P; short version). SCAS-P measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety, and specific fears). This yields a minimum possible score of 0 and a maximum possible score of 24. Higher scores indicate greater severity of symptoms.
Change from baseline children's reported psychological adjustment to immediately after the intervention | baseline and immediately after the intervention
  Measured by Strengths and Difficulties Questionnaire Child Report (SDQ). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximum value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.
Change from baseline parent-reported psychological adjustment to immediately after the intervention | baseline and immediately after the intervention
  Measured by Strengths and Difficulties Questionnaire Parental Report (SDQ-P). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximum value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.
Children's reported psychological adjustment at 1 year | 1 year after the intervention
  Measured by Strengths and Difficulties Questionnaire Child Report (SDQ). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximum value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.
Parent-reported psychological adjustment at 1 year | 1 year after the intervention
  Measured by Strengths and Difficulties Questionnaire Parental Report (SDQ-P). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximum value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.

SECONDARY OUTCOMES:
Change from baseline self-concept to immediately after the intervention | baseline and immediately after the intervention
  Measured by the Self-Concept Form 5 (AF-5). It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Children's self-concept at 1 year | 1 year after the intervention
  Measured by the Self-Concept Form 5 (AF-5). It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Change from baseline social worries to immediately after the intervention | baseline and immediately after the intervention
  Measured by the Social Worries Questionnaire for pupils (SWQ-PU). It evaluates children's worries in different social situations. In general, the higher the score, the more severe the symptomatology.
Children's social worries at 1 year | 1 year after the intervention
  Measured by the Social Worries Questionnaire for pupils (SWQ-PU). It evaluates children's worries in different social situations. In general, the higher the score, the more severe the symptomatology.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Melero, PhD, Principal Investigator — Universidad Miguel Hernández de Elche; Mireia Orgilés, Professor, Study Director — Universidad Miguel Hernández de Elche; José Pedro Espada, Professor, Study Director — Universidad Miguel Hernández de Elche
Locations (1):
- Universidad Miguel Hernández de Elche, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Starting after finishing all analysis and publication
Access Criteria: Upon request and verification by the principal investigator to consult the available data. The use of the data for distribution in any format is not permitted.

REFERENCES:
- [Background] Essau, C. A., & Ollendick, T. H. (2013). The Super Skills for Life Programme. London, Reino Unido: University of Roehampton
- [Background] Essau CA, Olaya B, Sasagawa S, Pithia J, Bray D, Ollendick TH. Integrating video-feedback and cognitive preparation, social skills training and behavioural activation in a cognitive behavioural therapy in the treatment of childhood anxiety. J Affect Disord. 2014;167:261-7. doi: 10.1016/j.jad.2014.05.056. Epub 2014 Jun 4. PMID 24999861
- [Background] Essau CA, Sasagawa S, Jones G, Fernandes B, Ollendick TH. Evaluating the real-world effectiveness of a cognitive behavior therapy-based transdiagnostic program for emotional problems in children in a regular school setting. J Affect Disord. 2019 Jun 15;253:357-365. doi: 10.1016/j.jad.2019.04.036. Epub 2019 Apr 16. PMID 31078836
- [Background] Fernández-Martínez, I., Espada, J. P., & Orgilés, M. (2019). Super Skills for Life: Eficacia de un programa transdiagnóstico de prevención indicada para los problemas emocionales infantiles. Revista de Psicología Clínica con Niños y Adolescentes, 6(3), 24-31. https://doi.org/10.21134/rpcna.2019.06.3.3
- [Background] Orgiles M, Fernandez-Martinez I, Espada JP, Morales A. Spanish version of Super Skills for Life: short- and long-term impact of a transdiagnostic prevention protocol targeting childhood anxiety and depression. Anxiety Stress Coping. 2019 Nov;32(6):694-710. doi: 10.1080/10615806.2019.1645836. Epub 2019 Jul 23. PMID 31334667
- [Background] Fernandez-Martinez I, Morales A, Espada JP, Essau CA, Orgiles M. Effectiveness of the program Super Skills For Life in reducing symptoms of anxiety and depression in young Spanish children. Psicothema. 2019 Aug;31(3):298-304. doi: 10.7334/psicothema2018.336. PMID 31292045
- [Background] Fernandez-Martinez I, Orgiles M, Morales A, Espada JP, Essau CA. One-Year follow-up effects of a cognitive behavior therapy-based transdiagnostic program for emotional problems in young children: A school-based cluster-randomized controlled trial. J Affect Disord. 2020 Feb 1;262:258-266. doi: 10.1016/j.jad.2019.11.002. Epub 2019 Nov 4. PMID 31733917
- [Background] Diego-Castaño, S., Prieto-Moya, J., Hermosín, N., & Orgilés, M. (2019). Eficacia del programa Super Skills en población clínica: un estudio piloto. 5 Congreso International de Psicología Clinica y Salud con Niños y Adolescentes, Oviedo, Spain. ISSN: 2695-4664
- [Background] Melero, S., Morales, A., & Orgilés, M. (2019, noviembre). Eficacia de la aplicación individual del programa Super Skills for Life para reducir síntomas emocionales en menores. 5 Congreso International de Psicología Clinica y Salud con Niños y Adolescentes, Oviedo, Spain. ISSN: 2695-4664
- [Background] Fernandez-Martinez I, Morales A, Espada JP, Orgiles M. Effects of Super Skills for Life on the social skills of anxious children through video analysis. Psicothema. 2020 May;32(2):229-236. doi: 10.7334/psicothema2019.240. PMID 32249749
- [Background] Orgiles M, Melero S, Fernandez-Martinez I, Espada JP, Morales A. Effectiveness of Video-Feedback with Cognitive Preparation in Improving Social Performance and Anxiety through Super Skills for Life Programme Implemented in a School Setting. Int J Environ Res Public Health. 2020 Apr 18;17(8):2805. doi: 10.3390/ijerph17082805. PMID 32325756
- [Background] Orgilés, M., Garrigós, E., Espada, J. P., & Morales, A. (2020). How does a CBT-based transdiagnostic program for separation anxiety symptoms work in children?: Effects of Super Skills for Life. Revista de Psicología Clínica con Niños y Adolescentes, 7(2), 9-15. https://doi.org/10.21134/rpcna.2020.07.2.1
- [Background] Orgilés, M., Espada, J. P, & Morales, A. (2020). How Super Skills for Life may help children to cope with the COVID-19: Psychological impact and coping styles after the program. Revista de Psicología Clínica con Niños y Adolescentes, 7(3), 88-93. https://doi.org/10.21134/rpcna.2020.mon.2048
- [Background] Melero, S., Orgilés, M., Fernández-Martínez, I., Espada, J. P., & Morales, A. (2021). Influence of implementation fidelity on the effectiveness of a CBT programme targeted emotional problems in childhood. Studies in Educational Evaluation, 68, 100975. https://doi.org/10.1016/j.stueduc.2021.100975
- [Background] Fernandez-Martinez I, Orgiles M, Espada JP, Essau CA, Morales A. Effects as a function of implementation fidelity of a transdiagnostic prevention program in young school-aged children. Eval Program Plann. 2021 Dec;89:102011. doi: 10.1016/j.evalprogplan.2021.102011. Epub 2021 Sep 16. PMID 34562670
- [Background] Melero S, Morales A, Espada JP, Orgiles M. Improving Social Performance Through Video-feedback with Cognitive Preparation in Children with Emotional Problems. Behav Modif. 2022 Jul;46(4):755-781. doi: 10.1177/0145445521991098. Epub 2021 Jan 29. PMID 33511861
- [Background] Melero S, Orgiles M, Espada JP, Morales A. Spanish version of Super Skills for Life in individual modality: Improvement of children's emotional well-being from a transdiagnostic approach. J Clin Psychol. 2021 Oct;77(10):2187-2202. doi: 10.1002/jclp.23148. Epub 2021 Apr 21. PMID 33882156
- [Background] Melero S, Morales A, Espada JP, Mendez X, Orgiles M. Effectiveness of Group vs. Individual Therapy to Decrease Peer Problems and Increase Prosociality in Children. Int J Environ Res Public Health. 2021 Apr 9;18(8):3950. doi: 10.3390/ijerph18083950. PMID 33918640
- See also: Description University of Roehampton research for Super Skills for Life program — https://www.superskillsforlife.com/